CLINICAL TRIAL: NCT07118293
Title: Developing and Examine the Efficacy of the Family-Centered Multi-Sensory Environment Intervention on Parent's Empowerment and Children's Engagement (MSE-PEACE) in Children With Developmental Disabilities and Their Parents: A Mixed Methods Study
Acronym: MSE-PEACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ling-Yi Lin, Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B-BR-113-022
Record Dates: First submitted 2025-06-13; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Developmental Disability
Keywords: Developmental Disabilities; Family-Centered Intervention; Multi-Sensory Environment; Parent Empowerment; Occupational Therapy; Child Engagement; Mixed Methods
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSE-PEACE Group (Experimental): Participants in this arm will receive the MSE-PEACE intervention, a family-centered multi-sensory environment program designed for children with developmental disabilities and their caregivers. The intervention includes 10 sessions delivered every 2 weeks, with each session lasting approximately 60 minutes. Sessions take place in a specialized sensory therapy room and are guided by certified occupational therapists.
  The intervention combines sensory-based activities with active parent-child co-participation. Each session is tailored to the child's sensory profile and developmental needs. Parents are engaged in goal-setting, activity participation, and follow-up support, including suggestions for home-based sensory activities and environmental adaptations. The program aims to improve children's functional engagement and emotional regulation, while enhancing caregiver empowerment, parenting competence, and family well-being.
  Interventions: Behavioral: MSE-PEACE

INTERVENTIONS:
Behavioral: MSE-PEACE — The MSE-PEACE (Multi-Sensory Environment-Parent Empowerment and Child Engagement) intervention is a family-centered, therapist-guided sensory integration program specifically developed for children with developmental disabilities and their caregivers. Unlike traditional child-only sensory therapies, this intervention actively involves parents in all stages-assessment, goal setting, activity participation, and follow-up.
  Each participant dyad (parent and child) attends 10 biweekly sessions (60 minutes each) in a structured sensory therapy space equipped with adjustable lighting, tactile materials, auditory inputs, and other multisensory tools. The intervention is tailored to each child's sensory processing profile and emotional regulation needs, while promoting parent-child co-regulation, bonding, and collaborative engagement.
  Occupational therapists facilitate the sessions using individualized strategies to support child-led participation and empower parents with real-time coaching,

SUMMARY:
The goal of this clinical trial is to learn whether a family-centered multi-sensory environment (MSE-PEACE) can help children with developmental disabilities and support their parents. The main questions it aims to answer are:

Can the MSE-PEACE program improve children's participation and emotional self-regulation? Does it help parents feel more confident and empowered in their caregiving role?

Participants will include children ages 3 to 12 years and their parents. All children have been diagnosed with a developmental disability such as autism, ADHD, or cerebral palsy. Participants will:

Join 10 multi-sensory sessions, held every 2 weeks, each lasting about 60 minutes Complete questionnaires and interviews before and after the sessions Receive support and suggestions for using sensory-based activities at home

This study will collect both survey and interview data to understand how the program affects children's daily functioning and how it supports parents' confidence and well-being.

DETAILED DESCRIPTION:
This quasi-experimental, single-group pretest-posttest mixed methods study examines the efficacy of a family-centered multi-sensory environment (MSE-PEACE) intervention for families of children with developmental disabilities (DD). The study is conducted at a multi-sensory therapy facility under the guidance of licensed occupational therapists, and aims to promote children's engagement and emotional self-regulation while strengthening parental empowerment and caregiving confidence.

The intervention integrates principles of sensory integration therapy with a family-centered approach, emphasizing shared decision-making, parent-child co-participation, and individualized sensory needs. The target population includes 20 children aged 3 to 12 years diagnosed with DD (e.g., autism spectrum disorder, ADHD, cerebral palsy, developmental delay) and their caregivers.

The MSE-PEACE program consists of 10 biweekly, 60-minute sessions delivered in a specialized sensory environment (e.g., "White Room" and "Rainbow Room"). Each session is tailored through therapist-family collaboration to meet the child's sensory profile and developmental goals. Parents are actively involved in each session and receive ongoing guidance on home-based sensory play and environmental adaptations.

Quantitative data will be collected pre- and post-intervention using validated tools to assess child outcomes (e.g., sensory processing, emotional regulation, functional participation) and parent outcomes (e.g., empowerment, parenting competence, stress, and parent-child relationship quality). Tools include the Short Sensory Profile 2, Emotion Regulation Checklist, Family Empowerment Scale, Parenting Stress Index, Parenting Sense of Competence Scale, and Parent-Child Relationship Inventory.

Qualitative data will be collected via semi-structured interviews with parents before and after the intervention. These interviews aim to capture parent experiences, perceptions of empowerment, interaction with service providers, and views on co-participation in therapy.

Quantitative analysis will involve paired t-tests to assess pre-post differences. Qualitative data will be analyzed using thematic analysis and integrated with quantitative results via joint displays, following a convergent mixed methods design.

The study expects to generate evidence for a practical and replicable family-centered sensory intervention model and to inform future community-based and home-based service designs for children with developmental disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 12 years
* Diagnosed with a developmental disability (e.g., autism spectrum disorder, attention-deficit/hyperactivity disorder, cerebral palsy, global developmental delay)
* Able to attend 10 biweekly intervention sessions in person with a caregiver
* Caregiver is the primary caregiver and agrees to actively participate in all sessions
* Caregiver is able to complete written questionnaires in Chinese
* Caregiver provides informed consent

Exclusion Criteria:

* Child has significant physical or behavioral challenges that prevent safe participation in a multi-sensory therapy setting (e.g., uncontrollable aggression, high seizure risk)
* Caregiver has cognitive or psychiatric conditions that significantly limit the ability to participate in shared sessions or complete questionnaires

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pediatric Volitional Questionnaire (Chinese version) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Pediatric Volitional Questionnaire (PVQ), adapted from the Volitional Questionnaire, is used to assess a child's motivation and engagement in different environments. It consists of 14 observational items such as curiosity, task initiation, persistence, and problem solving. Each item is scored on a 4-point scale from "Passive" to "Spontaneous." The scores range from 14 to 56, higher scores mean better engagement. Observations are conducted during 15-30 minutes of free play in natural settings (e.g., therapy room, playground, or home). The PVQ has demonstrated strong reliability and validity in children with developmental delays, with an item separation reliability coefficient of 0.97. This study uses the PVQ to evaluate changes in children's volitional behavior and functional participation before and after the MSE-PEACE intervention.
Short Sensory Profile 2 - Chinese Version (SSP-2) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Short Sensory Profile 2 (SSP-2) is a 34-item caregiver-reported questionnaire used to evaluate sensory processing patterns in children aged 3 to 14 years. It assesses four sensory quadrants: sensory seeking, sensory avoiding, sensory sensitivity, and low registration (observer). Caregivers rate each item based on the child's typical behavior in daily life using a 5-point Likert scale (1 = Almost Never to 5 = Almost Always). Higher scores within each quadrant indicate greater difficulties in sensory processing according to age norms.
  The Chinese version of SSP-2 has been translated and validated in prior studies, showing strong internal consistency (Cronbach's α = 0.949). This study uses the SSP-2 to assess changes in children's sensory processing patterns before and after the MSE-PEACE intervention.
Emotion Regulation Checklist - Chinese Version (ERC) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Emotion Regulation Checklist (ERC) is a 24-item parent-report measure used to evaluate children's emotion regulation abilities. Parents rate how frequently their child demonstrates specific emotional behaviors in daily life using a 4-point Likert scale (1 = Never to 4 = Almost Always). The ERC includes two subscales: Emotion Regulation (ERC-ER), which reflects a child's ability to understand and express emotions appropriately, and Lability/Negativity (ERC-L/N), which reflects emotional dysregulation and instability. Higher ERC-ER scores indicate better emotion regulation, while higher ERC-L/N scores indicate greater emotional dysregulation.
  The Chinese version has shown acceptable internal consistency, with Cronbach's α values of 0.88 (ERC-ER) and 0.64 (ERC-L/N). This study uses the ERC to assess changes in children's emotional self-regulation following the MSE-PEACE intervention.
Family Empowerment Scale - Chinese Version (FES) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Family Empowerment Scale (FES) is a 34-item self-report questionnaire designed to measure caregivers' perceptions of their empowerment when raising a child with disabilities. It evaluates empowerment across three domains: Family (12 items), Service System (12 items), and Community/Political (10 items). Respondents rate items using a 6-point Likert scale from 0 ("Not applicable") to 5 ("Very often"), with higher scores indicating higher levels of perceived empowerment.
  The Chinese version used in this study was translated using a forward-backward translation process, reviewed by an expert panel, and pre-tested with caregivers for clarity and cultural relevance. The original FES demonstrates strong psychometric properties, including internal consistency reliability coefficients of 0.88, 0.87, and 0.88 across the three subscales, and test-retest reliabilities of 0.83, 0.77, and 0.85, respectively.
Parenting Sense of Competence Scale - Chinese Version (PSOC) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Parenting Sense of Competence Scale - Chinese Version (PSOC) is a 17-item self-report questionnaire used to assess parents' perceptions of their competence in the parenting role. The scale includes two subscales: (1) Parenting Efficacy (skills and knowledge) and (2) Parenting Satisfaction (comfort and value). Responses are rated on a Likert scale from 1 to 6, higher scores reflect better sense of competence that parents feel about their caregiving.
  The Chinese version of the PSOC has demonstrated good psychometric properties, including internal consistency (Cronbach's α = .85) and test-retest reliability (intraclass correlation coefficient = .87). It also shows construct validity through correlations with measures of self-esteem and postpartum depression.
  This study uses the PSOC to evaluate changes in parenting confidence and satisfaction following participation in the MSE-PEACE intervention.
Parenting Stress Index - Fourth Edition Short Form (Chinese Version) (PSI-4-SF) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Parenting Stress Index, Fourth Edition Short Form (Chinese Version) (PSI-4-SF) is a 36-item self-report questionnaire used to assess the level and sources of stress parents experience in their caregiving role. It includes three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The tool helps identify whether parenting stress stems from parent characteristics, child characteristics, or the relationship between parent and child. Higher scores reflected a greater sense of stress in parenting.
  The Chinese version used in this study demonstrated strong psychometric properties, with internal consistency coefficients ranging from 0.92 to 0.95 across subscales and 0.97 for the total scale. Factor analysis supported the consistency of the translated scale structure with the original.
  This study uses the PSI-4-SF to examine changes in parenting stress levels and contributing factors before and after the MSE-PEACE.

SECONDARY OUTCOMES:
Parent-Child Relationship Inventory - Chinese Version (PCRI) | At baseline (within 1 week before the first intervention session) and immediately after completion of the 10th session (within 1 week)
  The Parent-Child Relationship Inventory (PCRI) is a 78-item parent-report questionnaire designed to assess the quality of the parent's relationship with their child. Items are rated on a 4-point Likert scale from "Strongly Agree" to "Strongly Disagree," including some reverse-scored items. The scale consists of seven subscales: Support, Satisfaction, Involvement, Communication, Limit Setting, Autonomy, and Role Orientation. Higher scores indicate a more positive perceived parent-child relationship.
  The Chinese version of the PCRI was translated and back-translated by bilingual professionals and reviewed by experts in occupational therapy to ensure conceptual and linguistic equivalence. It was pilot-tested with caregivers of children aged 3 to 6 to ensure clarity and cultural relevance. Internal consistency ranges from 0.59 to 0.82 across subscales, with acceptable reliability for most dimensions.
Therapy Attitude Inventory - Chinese Version (TAI) | At immediately after completion of the 10th session (within 1 week)
  The Therapy Attitude Inventory - Chinese Version (TAI) is a 10-item self-report questionnaire designed to measure caregiver satisfaction with child-focused therapeutic interventions. Respondents rate their perceptions of treatment helpfulness and satisfaction. Higher scores means a greater sense of helpfulness and satisfaction. The TAI has demonstrated strong internal consistency (Cronbach's α = 0.91) and four-month test-retest reliability (r = 0.85).
  The Chinese version of the TAI was translated and culturally adapted by the research team in previous studies. In this study, it will be administered to parents immediately following the intervention to assess overall satisfaction with the MSE-PEACE program. The questionnaire takes approximately 5 to 10 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy, National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared publicly due to the sensitive nature of the data involving young children with developmental disabilities and their families. Data privacy and confidentiality cannot be sufficiently protected for public sharing.

REFERENCES:
- [Background] Zablotsky B, Black LI, Maenner MJ, Schieve LA, Danielson ML, Bitsko RH, Blumberg SJ, Kogan MD, Boyle CA. Prevalence and Trends of Developmental Disabilities among Children in the United States: 2009-2017. Pediatrics. 2019 Oct;144(4):e20190811. doi: 10.1542/peds.2019-0811. PMID 31558576
- [Background] Unwin KL, Powell G, Price A, Jones CR. Patterns of equipment use for autistic children in multi-sensory environments: Time spent with sensory equipment varies by sensory profile and intellectual ability. Autism. 2024 Mar;28(3):644-655. doi: 10.1177/13623613231180266. Epub 2023 Jul 7. PMID 37421130
- [Background] Novakovic N, Milovancevic MP, Dejanovic SD, Aleksic B. Effects of Snoezelen-Multisensory environment on CARS scale in adolescents and adults with autism spectrum disorder. Res Dev Disabil. 2019 Jun;89:51-58. doi: 10.1016/j.ridd.2019.03.007. Epub 2019 Mar 29. PMID 30933867
- [Background] DeChillo N, Koren PE, Schultze KH. From paternalism to partnership: family and professional collaboration in children's mental health. Am J Orthopsychiatry. 1994 Oct;64(4):564-76. doi: 10.1037/h0079572. PMID 7847572
- [Background] Hotz GA, Castelblanco A, Lara IM, Weiss AD, Duncan R, Kuluz JW. Snoezelen: a controlled multi-sensory stimulation therapy for children recovering from severe brain injury. Brain Inj. 2006 Jul;20(8):879-88. doi: 10.1080/02699050600832635. PMID 17046800
- [Background] Dwamena F, Holmes-Rovner M, Gaulden CM, Jorgenson S, Sadigh G, Sikorskii A, Lewin S, Smith RC, Coffey J, Olomu A. Interventions for providers to promote a patient-centred approach in clinical consultations. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD003267. doi: 10.1002/14651858.CD003267.pub2. PMID 23235595